CLINICAL TRIAL: NCT01566994
Title: Comparing Population Cessation Services With Emphasis on Unmotivated Smokers
Brief Title: Comparing Population Cessation Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Responsible Party: Principal Investigator, James O. Prochaska, Professor, University of Rhode Island
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: DA022291
Record Dates: First submitted 2012-01-31; First posted 2012-03-30 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Cancer
Keywords: smoking cessation
MeSH Terms: conditions — Neoplasms; Smoking Cessation | interventions — Motivational Interviewing; Combined Modality Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TTM Tailored (Experimental)
  Interventions: Behavioral: TTM Tailored
- Motivational Enhancement Therapy (Experimental)
  Interventions: Behavioral: Motivational Enhancement Therapy
- Integrated Treatment (Experimental)
  Interventions: Behavioral: Integrated Treatment

INTERVENTIONS:
Behavioral: TTM Tailored — This treatment is tailored on three occasions (baseline, 6, and 24 weeks) on each of the 14 TTM variables. This treatment provides both normative and ipsative feedback on each of the variables found to predict progress across specific stages
  Other Names: TTM Expert System
  Arms: TTM Tailored
Behavioral: Motivational Enhancement Therapy — This intervention will be driven by the manual developed by Carpenter et al. (2004) based on the USPHS recommendations for smokers not motivated to quit and for those who become ready to set a quit date.
  Other Names: MET
  Arms: Motivational Enhancement Therapy
Behavioral: Integrated Treatment — This enhanced condition would combine MET, Reduction Counseling and NRT and TTM Tailoring.
  Other Names: Combined treatment
  Arms: Integrated Treatment

SUMMARY:
If the treatment combining Motivation Enhancement, Reduction Counseling, Nicotine Replacement Therapy and Transtheoretical tailored interventions produces an increasing treatment trajectory, it will produce unprecedented impacts with unmotivated smokers specifically and population cessation generally. These recruitment and intervention strategies require limited resources from health care providers and could be readily disseminable to other health care systems for application with populations of smokers, especially unmotivated smokers who have been understudied and underserved.

DETAILED DESCRIPTION:
This proposal addresses major gaps in research for nicotine addiction treatments for entire populations of smokers and for the 80% who are not motivated to quit. Nicotine addiction is just like other drug addictions in terms of breaking the addiction cycle. Researchers and providers differ on whether treatment emphasis should be on clinician-based counseling, biologically-based medications, computer-based tailored communications or a combination of these. There is a lack of comparative research on population treatments to compare effectiveness, cost-effectiveness and enhancement of quality of life. Such comparative research would provide health care systems and providers with evidence on how to best serve entire populations of smokers, especially unmotivated smokers who are seriously underserved. This research will compare the four most highly recommended treatments: 1. Motivation Enhancement Therapy (MET) plus NRT; 2.Tailored communications based on the Transtheoretical Model (TTM), and 3. The combination of these treatments.

ELIGIBILITY:
Inclusion Criteria:

* smoker

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2500 (Actual)
Dates: Start 2010-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Smoking cessation (quit) rate | 24 months
  Self-report point prevalence abstinence

CONTACTS AND LOCATIONS:
Overall Officials: James O Prochaska, Ph.D., Principal Investigator — Univeristy of Rhode Island
Locations (1):
- University of Rhode Island, Kingston, Rhode Island, United States